CLINICAL TRIAL: NCT06900504
Title: "The Effect of Sleep Hygiene Training Given to Heart Failure Patients on Their HospitalAcquired Insomnia Level": Randomized Controlled Trial
Brief Title: "The Effect of Sleep Hygiene Training Given to Heart Failure Patients on Their HospitalAcquired Insomnia Level"
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: muş alp
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Sleep hygiene education will be given to the experimental group.
  Interventions: Other: Sleep hygiene education
- Control Group (No Intervention): Standard application procedure will be applied to the control group.

INTERVENTIONS:
Other: Sleep hygiene education — A structured training booklet will be prepared to ensure sleep hygiene for individuals. In addition, sleep hygiene training will be provided to individuals.
  Arms: Experimental Group

SUMMARY:
The purpose of this study is to examine the effect of sleep hygiene education given to heart failure patients on the level of hospital-acquired insomnia of the patients. Participants will be randomly assigned to groups as experimental and control groups. Standard application procedure will be applied to the control group. Sleep hygiene education will be given to the experimental group.

Research Hypotheses H0: Sleep hygiene education given to heart failure patients does not have a positive effect on the level of hospital-acquired insomnia of the patients.

H1: Sleep hygiene education given to heart failure patients has a positive effect on the level of hospital-acquired insomnia of the patients.

DETAILED DESCRIPTION:
Heart failure (HF) is a life-threatening health problem. HF is considered a public health burden when the incidence, prevalence, healthcare expenditures, morbidity, mortality and poor quality of life are considered. Heart failure is prevalent in 6.5 million people in the United States, approximately 900,000 people are discharged from the hospital and more than 78,000 people die each year. HF, which has a high mortality and morbidity rate, has many symptoms. HF patients experience various physical and emotional complaints such as dyspnea, fatigue, edema, sleep disorders, depression and chest pain. Pharmacological and non-pharmacological treatment methods are used to improve sleep quality in chronic diseases. However, the inadequacy of pharmacological treatment methods and the fact that they cause various problems have brought non-pharmacological treatment methods to the forefront. One of the most frequently used methods in the non-pharmacological treatment of sleep problems is sleep hygiene training. The concept of sleep hygiene was first used by Peter Hauri. Sleep hygiene aims to provide behaviors that will ensure good sleep by avoiding individual behaviors that disrupt normal sleep patterns. The purpose of this study is to examine the effect of sleep hygiene education given to heart failure patients on the level of hospital-acquired insomnia of the patients. Participants will be randomly assigned to groups as experimental and control groups. Standard application procedure will be applied to the control group. Sleep hygiene education will be given to the experimental group.

Research Hypotheses H0: Sleep hygiene education given to heart failure patients does not have a positive effect on the level of hospital-acquired insomnia of the patients.

H1: Sleep hygiene education given to heart failure patients has a positive effect on the level of hospital-acquired insomnia of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Being literate
* Being a heart failure patient
* Being hospitalized for at least 1 week and staying for another week
* Not having a condition that prevents verbal communication
* Not having a diagnosed psychiatric problem
* Being a volunteer to participate in the research

Exclusion Criteria:

* Having a verbal communication disability
* Having a diagnosed psychiatric problem

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Hospital-acquired insomnia | 1 months
  Insomnia Score Average

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University Research Hospital, Erzurum, Turkey (Türkiye)